CLINICAL TRIAL: NCT02898727
Title: A Phase II Study of Local Therapy Only (Stereotactic Radiosurgery and/or Surgery) for Treatment of up to 5 Brain Metastases From HER2 Positive Breast Cancer
Brief Title: A Study of Local Therapy for the Treatment of Brain Metastases From HER2 Positive Breast Cancer
Acronym: Local HER-O
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROG 16.02
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Hyperthermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Local Therapy (Other): The local therapy offered will be determined by the participant's doctor in consultation with the site multidisciplinary team and will be dependent on the size and location of the brain metastases.
  Neurosurgery: The surgery may be performed up to 6 weeks before participant being registered on the trial or up to 4 weeks after registration.
  Sometimes stereotactic radiosurgery is required to be delivered to the cavity left after the metastasis has been removed (Cavity Boost).
  Stereotactic Radiosurgery: Treatment is to commence within 4 weeks of study registration. The size, number and location of the brain metastasis will determine the dose and fractionation schedule of radiotherapy.
  Interventions: Other: Local Therapy

INTERVENTIONS:
Other: Local Therapy — Neurosurgery: The decision whether or not to recommend neurosurgery will be made independently of this research study. The complexity and length of the surgery depends on the size and location of the tumour(s).
  Stereotactic Radiosurgery: If the participant will be receiving stereotactic radiosurgery (either alone or in combination with neurosurgery), the Radiation Oncologist will organise for the participant to have a Radiotherapy planning. Single metastasis, smaller than or equal to 2cm, may require 1 fraction. Alternately, multiple metastasis, metastasis in the brain stem, or those bigger than 2cm will required multiple fractions to treat. The dose range for the study is 20Gy/1 fraction to 24Gy/3 fractions.

SUMMARY:
This study aims to show that brain metastases from Human Epidermal Growth Factor Receptor Type 2 (HER2) positive breast cancers are able to be controlled by local therapies, Stereotactic Radiosurgery (SRS) and/or Neurosurgery (NS), without the need for Whole Brain Radiotherapy (WBRT).

DETAILED DESCRIPTION:
For patients who have Human Epidermal Growth Factor Receptor Type 2 (HER2) positive breast cancer, which has metastasised to the brain, the main treatment options for these brain metastases are Whole Brain Radiotherapy (WBRT), Stereotactic Radiosurgery (SRS) and Neurosurgery (NS).

The purpose of the study is to determine:

1. . How likely the tumours are controlled after treatment with local therapies Neurosurgery (NS) and/or Stereotactic Radiosurgery (SRS).
2. . How likely is it that other tumours develop at new sites in the brain when no Whole Brain Radiotherapy (WBRT) is given.

This study is aiming to recruit 50 participants that have HER2 positive metastatic breast cancer with 1-5 synchronous brain metastases, with at least one metastasis requiring treatment.

The local treatment offered will be determined by the participant's doctor in consultation with the site multidisciplinary team and will be dependent on the size and location of the brain metastases. Each treatment will be performed by the specialist in that field, i.e. neurosurgeon and/or radiation oncologist.

Neurosurgery: The decision whether or not to recommend neurosurgery will be made independently of this research study. The surgery may be performed up to 6 weeks before participant being registered on the trial or up to 4 weeks after registration. The complexity and length of the surgery depends on the size and location of the tumour(s).

Sometimes stereotactic radiosurgery is required to be delivered to the cavity left after the metastasis has been removed (also known as a cavity boost). Timing of Cavity SRS is at the discretion of the treating team. SRS cavity boost must be given after registration and can be given up to 8 weeks after NS resection.

Stereotactic Radiosurgery: If the participant will be receiving stereotactic radiosurgery (either alone or in combination with neurosurgery), the Radiation Oncologist will organise for the participant to have a Radiotherapy planning. Treatment is to commence within 4 weeks of study registration.

The size, number and location of the brain metastasis will determine the dose and fractionation schedule of radiotherapy. Single metastasis, smaller than or equal to 2cm, may require 1 fraction. Alternately, multiple metastasis, metastasis in the brain stem, or those bigger than 2cm will required multiple fractions to treat. The dose range for the study is 20Gy/1 fraction to 24Gy/3 fractions. Each fraction is given on a separate day.

All participants will be followed up at 3 monthly intervals for 12 months after completing their trial treatment (i.e. from the day of their last SRS treatment or neurosurgery, the latter of the two).

At each follow-up visit they will have a clinic visit with the study doctor who to assess any symptoms, record current medications and/or surgeries, monitor their brain metastasis, have a blood test and imaging (CT scan, bone scan and MRI brain).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Metastatic HER2 positive breast cancer
* 1-5 synchronous brain metastases
* At least one metastases requiring treatment
* Maximum volume of any single PTV <10cm3
* Summated volume of all lesions to be treated with SRS is < 15cm3. If a lesion is too small for treatment and will be observed, then its volume is not included in this summation
* ECOG 0-2
* Absent or stable extracranial disease or active extracranial disease that is likely to be controlled with further HER-2 targeted therapy
* Receiving systemic HER2 targeted therapy, or planned to receive within 4 weeks of completion of brain metastasis treatment
* Able to undergo MRI scanning

Exclusion Criteria:

* Previous treatment to the target brain metastases (excluding surgery within 6 weeks of registration)
* Previous whole brain radiotherapy (WBRT)
* Any brain metastasis that is greater than 30mm in size and unable to be resected
* Leptomeningeal disease
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
to assess the percentage of patients treated with whole brain radiotherapy within 12 months after completion of local therapy | 12 months after completion of local therapy

SECONDARY OUTCOMES:
To describe distant brain failure incidence (overall and by number of treated metastases) | 12 months after completion of local therapy
To describe local brain failure incidence, at any site of SRS or surgery | 12 months after completion of local therapy
To describe extra-cranial failure incidence | 12 months after completion of local therapy
To describe the pattern of first failure | 12 months after completion of local therapy
To describe overall survival and cause of death (neurologic vs. non-neurologic) | 12 months after completion of local therapy
To describe adverse events and need for corticosteroids | Baseline and at 7-14 days, 3 months, 6 months, 9 months, and 12 months after completion of local therapy
To describe neurocognitive function using the mini-mental state examination (MMSE) | Baseline, and at 3, 6, 9, and 12 months after completion of local therapy

CONTACTS AND LOCATIONS:
Overall Officials: Claire Phillips, Dr, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia